CLINICAL TRIAL: NCT06583720
Title: Comparative Study Between Photodynamic Therapy with LED Associated with Probiotics in the Treatment of Halitosis - Controlled Randomized Clinical Trial
Brief Title: Comparative Study Between Photodynamic Therapy with LED Associated with Probiotics in the Treatment of Halitosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaliFAPESP
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Experimental): Participants in this group will perform brushing, dental floss and tongue scraper.
  Interventions: Procedure: Oral hygiene at home
- aPDT group (Experimental): Participants in this group will receive brushing, dental floss, tongue scraper and aPDT with blue LED and annatto.
  Interventions: Procedure: Oral hygiene at home; Procedure: aPDT
- aPDT and Probiotics group (Experimental): Participants in this group will receive brushing, dental floss, lingual scraper and aPDT with blue LED, annatto and probiotic lozenges containing Streptococcus salivarius K12 (BLIS K12®).
  Interventions: Procedure: Oral hygiene at home; Procedure: aPDT; Dietary Supplement: Probiotics
- Probiotics group (Experimental): Participants in this group will receive brushing, dental floss, lingual scraper and probiotic lozenges containing Streptococcus salivarius K12 (BLIS K12®).
  Interventions: Procedure: Oral hygiene at home; Dietary Supplement: Probiotics

INTERVENTIONS:
Procedure: Oral hygiene at home — Participant will be taught on how to correctly brush their teeth, use dental floss and scrape their tongues at home.
Procedure: aPDT — A weekly aPDT session will be performed for a period of 30 days, with the photosensitizer (PS) annatto manipulated at a concentration of 20% (Fórmula e Ação®). 2 ml (quantity measured with a pipette) will be applied to the middle third and dorsum of the tongue for 2 minutes for incubation (pre-irradiation time). The excess will be removed with a suction device in order to keep the surface moist with the PS itself. Six points will be irradiated with a distance of 1 cm between them, considering the light scattering halo; the LED will be positioned at a distance from the tongue so as to form a 2 cm halo at each point. The device will be previously calibrated with a wavelength of 395-480 nm, for 20 seconds per point, energy of 9.6 J.
  Arms: aPDT and Probiotics group; aPDT group
Dietary Supplement: Probiotics — Probiotic lozenges containing Streptococcus salivarius K12 (BLIS K12®) (OralBiotic; Master Products, Fort Lauderdale, Florida, United States) will be used. Each patient will receive 60 lozenges, which should be allowed to dissolve slowly and completely in the mouth. Patients are instructed to use the lozenges twice a day for a period of 30 days.
  Arms: Probiotics group; aPDT and Probiotics group

SUMMARY:
Halitosis is a term that defines any odor or bad smell coming from the oral cavity, which can have a local or systemic origin. This project aims to verify if there is a difference in the effectiveness of treatment with antimicrobial photodynamic therapy (aPDT) with LED associated with treatment using probiotics in reducing halitosis. 92 participants, aged 18 to 60 years, diagnosed with halitosis, presenting sulfhydride (SH2) ≥ 112 ppb in gas chromatography will be selected. Participants will be randomly divided into 4 groups (n=23), which will receive different treatments: Group 1 (control): brushing, dental floss and tongue scraper; Group 2: brushing, dental floss, tongue scraper and aPDT with blue LED and annatto; Group 3: brushing, dental flossing, tongue scraper and aPDT with blue LED, annatto and probiotic lozenges containing Streptococcus salivarius K12 (BLIS K12®); Group 4: brushing, dental flossing, tongue scraper and probiotic lozenges containing Streptococcus salivarius K12 (BLIS K12®). The results of the halimetry will be compared before, immediately after the treatments, thirty days after and sixty days after. The microbiological analysis will be performed by counting the colony forming unit of viable bacteria in the tongue coating at these same times. The microbiome analysis will be performed before, thirty days after and sixty days after the treatments after DNA extraction. All groups will be treated with oral hygiene instructions with a toothbrush, toothpaste and dental floss as well as receiving material for this practice. The normality of the data will be measured by the Shapiro-Wilk test, and in the case of normality the Analysis of Variance (ANOVA) test will be applied, and in the case of non-parametric data, the Kruskal-Wallis test will be used. The Wilcoxon test will be used to analyze the results of each treatment in the two study periods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of halitosis showing sulfhydride (SH2) ≥ 112 ppb in gas chromatography.

Exclusion Criteria:

* Individuals with dentofacial anomalies (such as cleft lip, cleft palate and nasopalatine);
* Undergoing orthodontic and/or orthopedic treatment;
* Undergoing oncological treatment;
* With systemic alterations (gastrointestinal, renal, hepatic)
* Undergoing antibiotic treatment up to 1 month before the research;
* Pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Halimetry Levels | Baseline, immediately after treatment, 30 days after treatment and 60 days after treatment.
  The collection of oral air will follow the manufacturer's instructions (Oral ChromaTM Manual Instruction), where the participant will be instructed to rinse with cysteine (10 mM) for 1 minute, then keep their mouth closed for another minute. A syringe from the same manufacturer, suitable for collecting oral air, will be placed in the patient's mouth. For 1 minute, the patient will remain with their mouth closed, breathing through their nose, without touching the syringe with their tongue. The plunger will be pulled out, we will empty the air from the syringe into the patient's mouth again and pull the plunger again to fill the syringe with the breath sample. We will clean the tip of the syringe with gauze to remove moisture from the saliva, place the gas injection needle on the syringe, and adjust the plunger to 0.5 ml. The collected gases are injected into the inlet port of the device with a single movement.

SECONDARY OUTCOMES:
Changes in Microbiological Analysis | Baseline, immediately after treatment, 30 days after treatment and 60 days after treatment.
  The samples will be collected with a swab on the back of the tongue, then placed in an eppendorf containing BHI (Brain Heart Infusion) serving as a transport medium, for later cultivation of these samples to be able to detect the total number of viable bacteria. Initially, the samples will be homogenized for 30 seconds in a Vortex apparatus, and then diluted in the order of 10-1 to 10-5 in a 96-well microtiter plate containing 180 microliters of PBS in each well. We take 20 microliters of each sample and follow the dilution sequence. After the dilution is performed, we will take 5 aliquots of 10 microliters of this suspension and they will be seeded in a petri dish with blood agar. The cultures will then be incubated for 72 hours at 37°C in an atmosphere of 85% nitrogen (N2), 10% carbon dioxide (CO2) and 5% hydrogen (H2), achieved through the use of an anaerobic generation system. This will provide visual access to the total number of viable bacteria in colony forming units (CFU).
Changes in Microbiome Analysis | Baseline, immediately after treatment, 30 days after treatment and 60 days after treatment.
  Tongue coating samples will be collected from the posterior third of the tongue using a sterile swab and deposited in 1.5 mL centrifuge tubes containing Tris-EDTA buffer (10 mM Tris-HCL, 0.1 mM EDTA, pH 7.5) and stored at -80 °C. After thawing, the samples will be vortexed for one minute. DNA extraction will be performed using the Master Pure DNA Extraction Kit (Epicentre Technologies Corp., Chicago, IL, USA) according to the manufacturer's instructions. The purified DNA will be resuspended in TE buffer. The microbiome and variations between communities will be analyzed using pyrosequencing and 16S rRNA gene metagenomics methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be added to OSF.
URL: https://osf.io/frk8w/?view_only=3de47176d5f241eb9bcaf3197da5581f

REFERENCES:
- [Derived] Mandetta ARH, Gallo JMAS, Ribeiro CDPV, Goncalves MLL, Sobral APT, Motta LJ, Horliana ACRT, Mesquita-Ferrari RA, Rodriguez VS, Prates RA, Duran CCG, Fernandes KPS, Bussadori SK. Comparative study of photodynamic therapy with LED and probiotics in the treatment of halitosis: protocol for a randomised controlled clinical trial. BMJ Open. 2025 Apr 25;15(4):e095544. doi: 10.1136/bmjopen-2024-095544. PMID 40280606